CLINICAL TRIAL: NCT04559230
Title: A Phase II, Multicenter, Prospective Study of Sacituzumab Govitecan in Recurrent Glioblastoma
Brief Title: Sacituzumab Govitecan in Recurrent Glioblastoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Principal Investigator, William Kelly, Clinical Investigator, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTMS# 20-0102; HSC20200576X (Other: UT Health Science Center San Antonio)
Record Dates: First submitted 2020-09-16; First posted 2020-09-22 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Recurrent Glioblastoma
Keywords: Trophoblast Cell-Surface Antigen 2; Trop-2; Sacituzumab Govitecan
MeSH Terms: conditions — Glioblastoma | interventions — sacituzumab govitecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Sacituzumab govitecan (Experimental): Dosing will be at 10 mg/kg on days 1 and 8 of a 21-day cycle
  Interventions: Drug: Sacituzumab Govitecan

INTERVENTIONS:
Drug: Sacituzumab Govitecan — Sacituzumab Govitecan will be administered by IV infusion over 3 hours for first administration and over 1 hour if tolerated. Subjects will be allowed to continue treatment until they have evidence of significant treatment-related toxicity or progressive disease.

SUMMARY:
This is an open-label single arm study. All patients will receive the study drug. The aim of the study is to compare overall survival (OS) of patients with recurrent brain tumor, known as Glioblastoma (GBM) having high levels of a protein, Trophoblast cell surface antigen 2 (Trop-2), expression on treatment with Sacituzumab Govitecan (SG) versus lomustine only which has been used in the past.

DETAILED DESCRIPTION:
Subjects are expected to participate for up to treatment duration with continued follow up for survival until one year after the last dose of study drug. The total duration of the active part of the study for each subject will be approximately 18 weeks, divided as follows:

* Up to 3 weeks predose (screening period)
* 3-week treatment periods of Sacituzumab govitecan
* Study termination visit 3-4 weeks after last dose of study medication

When a subject has completed the study termination or early termination visit, he/she and/or a family member will be contacted for survival information every 3 months until one year from last study dose.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age.
2. Ability to understand the purposes and risks of the study and has signed a written informed consent form approved by the investigator's IRB/Ethics Committee.
3. Histologically confirmed IDH wild type (primary) GBM. Molecular GBM (as per cIMPACT-NOW 3) is allowed as is gliosarcoma and epithelioid glioblastoma. IDH-mutant glioma is not allowed.
4. Progression following standard combined modality treatment with radiation and temozolomide chemotherapy if O6-Methylguanine-DNA Methyltransferase (MGMT) methylated.

   * Prior temozolomide is not required for MGMT unmethylated, but patient must have received standard doses of radiation.
   * Inclusion of additional investigational therapy with standard frontline therapy is not exclusionary. No additional lines of therapy given for recurrent disease.
   * Prior tumor-treating field therapy is not excluded, nor considered and additional line of therapy as this is often given concurrently with other therapy lines.
5. Patients may have had been operated for recurrence, but if operated must have had surgery a minimum of 2 weeks prior to enrollment and have an MRI completed within 48 hours following surgery.
6. No radiotherapy within the 3 months prior to the diagnosis of progression.
7. Willingness to forego tumor-treatment field (Optune) therapy during participation in the study.
8. Stable or decreasing dosage of steroids for 7 days prior to the baseline MRI scan.
9. Recovered from toxicities of prior therapy to grade 0 or 1, except for neuropathy (Grade ≤2) and alopecia.
10. ECOG performance status ≤ 2.
11. Life expectancy of at least 6 months.
12. Acceptable liver function:

    * Bilirubin ≤ 1.5 times upper limit of normal
    * AST (SGOT) and ALT (SGPT) ≤ 3.0 times upper limit of normal (ULN)
13. Acceptable renal function:

    • Creatinine clearance ≥30 mL/minute according to the Cockcroft and Gault formula
14. Acceptable hematologic status (without hematologic support):

    * ANC ≥1500 cells/uL
    * Platelet count ≥100,000/uL
    * Hemoglobin ≥9.0 g/dL
15. All women of childbearing potential must have a negative serum pregnancy test and male and female subjects must agree to use effective means of contraception (surgical sterilization or the use or barrier contraception with either a condom or diaphragm in conjunction with spermicidal gel or an IUD) with their partner from entry into the study through 6 months after the last dose.
16. Availability of biological material for central review and biomarker evaluation.
17. Untreated recurrent or residual disease that is measurable by RANO criteria at time of enrollment. Multifocal and infratentorial disease is allowed.
18. Positive Trop-2 expression (H-Score ≥200), as verified by central review at University of Texas Health Science Center at San Antonio (UTHSA).

Exclusion Criteria:

1. Prior treatment with bevacizumab or other VEGF inhibitors or VEGF-Receptor signaling inhibitors
2. The subject is receiving warfarin (or other coumarin derivatives) and is unable to switch to low molecular weight heparin (LMWH) before the first dose of study drug.

3 The subject has evidence of acute intracranial or intratumoral hemorrhage either by MRI or computerized tomography (CT) scan. Subjects with resolving hemorrhage changes, punctate hemorrhage, or hemosiderin are eligible.

4. The subject is unable to undergo MRI scan (eg, has pacemaker). 5. The subject has received enzyme-inducing anti-epileptic agents within 14 days of study drug (eg, carbamazepine, phenytoin, phenobarbital, primidone).

6. The subject is pregnant or breast-feeding. 7. The subject has serious intercurrent illness, such as:

* hypertension (two or more blood pressure [BP] readings performed at screening of > 150 mmHg systolic or > 100 mmHg diastolic) despite optimal treatment
* non-healing wound, ulcer, or bone fracture
* significant cardiac arrhythmias
* untreated hypothyroidism
* unhealed rectal or peri-rectal abscess
* uncontrolled active infection
* symptomatic congestive heart failure or unstable angina pectoris within 3 months prior study drug
* any history of cardiac arrhythmia or heart block
* stroke or transient ischemic attack within 6 months 8. The subject has received any of the following prior anticancer therapy:
* Non-standard radiation therapy such as brachytherapy, systemic radioisotope therapy (RIT), or intra-operative radiotherapy (IORT). Note: stereotactic radiosurgery (SRS) is allowed
* Systemic therapy (including investigational agents and small-molecule kinase inhibitors) or non-cytotoxic hormonal therapy (eg, tamoxifen) within 7 days or 5 half-lives, whichever is shorter, prior first dose of study drug
* Biologic agents (antibodies, immune modulators, vaccines, cytokines) within 21 days prior to first dose of study drug
* Nitrosoureas or mitomycin C within 42 days, or metronomic/protracted low-dose chemotherapy within 14 days, or other cytotoxic chemotherapy within 28 days, prior to first dose of study drug
* Prior treatment with carmustine wafers 9. Patients with radiographically or clinically apparent leptomeningeal involvement are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-01-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | 6 months
  Overall survival at 6 months including participants whose disease state has progressed

SECONDARY OUTCOMES:
Progression free survival (PFS) | 6 months
  To assess the progression-free survival (PFS) of these patients on SG vs historical control of lomustine monotherapy
Overall Response Rate (ORR) | 6 week intervals for 6 months, then every 3 months until End of Treatment ( defined as evidence of significant treatment related toxicity or progressive disease)
  To assess the Overall Response Rate (ORR) of these patients on SG by Response Assessment in Neuro-Oncology (RANO) criteria

CONTACTS AND LOCATIONS:
Overall Officials: William Kelly, MD, Principal Investigator — Mays Cancer Center, UT Health San Antonio
Locations (3):
- United States (3):
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Texas Oncology Austin, Austin, Texas
  - University of Texas Health Science Center San Antonio at the Cancer Therapy and Research Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No